CLINICAL TRIAL: NCT03317327
Title: REPORT; REirradiation and PD-1 Blockade On Recurrent Squamous Cell Head and Neck Tumors
Brief Title: REirradiation and Programmed Cell Death Protein 1 (PD-1) Blockade On Recurrent Squamous Cell Head and Neck Tumors
Acronym: REPORT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Åse Bratland, Principal Investigator, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-686_REPORT
Record Dates: First submitted 2017-09-25; First posted 2017-10-23 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: HNSCC; Nivolumab; immunotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Nivolumab; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Exploratory
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nivolumab (Experimental): Nivolumab, intravenous every 2nd week (1 cycle = 2 weeks), dose escalation schedule (1.0, 3.0 mg/kg), for a maximum of 12 months or until disease progression.
  Interventions: Drug: Nivolumab; Radiation: Radiotherapy (RT)

INTERVENTIONS:
Drug: Nivolumab — Nivolumab is a humanized antibody used in cancer immunotherapy.
  Other Names: Opdivo
Radiation: Radiotherapy (RT) — Radiotherapy (RT) will be given to a total dose of 60 Gy (1,5 Gy fractions twice daily) for a total period of 4 weeks

SUMMARY:
Each subject will participate in the trial until death, drop out, or loss-to follow-up from the time the subject signs the Informed Consent Form (ICF) through the final contact. After a screening phase of up to 28 days, each eligible subject will receive nivolumab. Two weeks after start of nivolumab the patients will receive radiotherapy (RT) to a total dose of 60 Gy, given as 1.5 Gy fractions twice daily for a total period of 4 weeks. Treatment with nivolumab will continue until disease progression, unacceptable adverse event(s), intercurrent illness that prevents further administration of treatment, Investigator's decision to withdraw the subject, noncompliance with trial treatment or procedures requirements, subject receives nivolumab for 12 months, pregnancy, or administrative reasons.

After the end of treatment, each subject will be followed for 30 days for adverse event monitoring serious adverse events (SAEs) will be collected for 90 days after the end of treatment. Patients without disease progression will have follow-up visits for 4 years after end of study therapy.

DETAILED DESCRIPTION:
In this study, the aim is to release the brake on the immune response by use of nivolumab, an inhibitory antibody against Programmed cell death protein 1 (PD-1). Nivolumab has shown efficacy and mild toxicity when given as monotherapy for HNSCC at a dose of 3.0 mg/kg every 2 weeks, which is the target dose in the present trial.

Radiotherapy is a powerful inducer of inflammation, and the expression of Programmed death-ligand 1 (PD-L1) is known to be enhanced by inflammatory cytokines, including interferon-gamma (IFNg). Experimental evidence from mice models have shown that radiotherapy induces increased PD-L1 expression in tumor tissue. Moreover, there is evidence suggesting that HNSCC with T-cell infiltration is more sensitive to radiotherapy. There is thus a strong rationale for combing PD-1 inhibitors with radiotherapy. However, this potential remains largely unexplored in humans. The investigators consider that head-and-neck cancer is a particularly attractive entity for investigating this therapeutic combination, because of i) the high radiosensitivity of this cancer form ii) the clinical efficacy of Programmed cell death protein 1 (PD-1) inhibitors as monotherapy in early clinical trials iii) the availability of tumor biopsies for translational/biomarker research.The RT given in the present study gives considerable side effects, related to inflammation that may be enhanced by Programmed cell death protein 1 (PD-1) blockade.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Recurrent or secondary primary squamous cell carcinoma originating from the oral cavity, oro/hypo-pharynx or larynx
* Prior radiotherapy (46-70Gy)
* Adequate newly obtained core or excisional biopsy of a recurrent tumor lesion
* Measurable disease
* Lesion available for biopsy during study treatment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of more than 12 months
* A minimum of 6 months since prior radiotherapy in the same area or minimum 4 weeks (28 days) since previous other cancer treatment
* Human papillomavirus positive and negative disease allowed
* Distant metastases allowed
* Adequate organ function based on clinical examination and lab values
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug
* Women must not be breastfeeding
* WOCBP should use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for a period of 90 days (duration of sperm turnover) plus the time required for the investigational drug to undergo five half-lives. The terminal half-life of nivolumab is up to 25 days

Exclusion Criteria:

* History of other prior malignancy, with the exception of curatively treated basal cell or squamous cell carcinoma of the skin, cervical cancer stage IB and stage I prostate cancer considered not necessary to treat
* Disease suitable for curative salvage surgery
* Treatment with any investigational medicinal product (IMP) that may interfere with the study treatment, within 4 weeks prior to first administration of study drug.
* Significant cardiac, pulmonary or other medical illness that would limit activity or survival
* Pregnancy or lactation.
* Known hypersensitivity to any of the components of the investigational product
* Patients who test positive for hepatitis B, C or HIV.
* Diagnosis of immunodeficiency or medical condition requiring systemic steroids or other forms of immunosuppressive therapy
* Autoimmune disease that has required systemic therapy within the past 2 years
* Any reason why, in the opinion of the investigator, the patient should not participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-09-09 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-11-28 (Actual)

PRIMARY OUTCOMES:
Incidence, nature, and severity of adverse events graded according to Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0. | 18 months (6 months after end of treatment)

SECONDARY OUTCOMES:
Progression-free survival (PFS) | After 12 months
  defined as the time from inclusion to the time of radiographic progression (as assessed by RECIST) or death from any cause during the study
Objective response rate (ORR) | 3 years
  defined as the proportion of patients with an objective tumor response
Overall survival (OS) | 5 years
  defined as the time from the date of inclusion to the date of death from any cause
Duration of response (DOR) | 3 years
  among patients with an objective response
Durable response rate (DRR) | 3 years
  defined as the proportion of patients with an objective tumor response lasting at least 6 months

OTHER OUTCOMES:
Immunological response | 3 years
  as assessed by gene profiling, immunohistochemistry, T cell assays, characterization of cell suspensions from tumor and peripheral blood
tumor evolution | 3 years
  as assessed by gene profiling, immunohistochemistry, characterization of cell suspensions from tumor and peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Åse Bratland, m, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT03317327/Prot_SAP_000.pdf